CLINICAL TRIAL: NCT00519324
Title: A Single Arm, Multi-center Phase II Study of RAD001 in Patients With Advanced Gastric Carcinoma Whose Cancer Has Progressed Despite Prior Treatment
Brief Title: Efficacy and Safety of Everolimus (RAD001) in Patients With Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C1201
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Advanced Gastric Cancer
Keywords: Gastric Cancer; RAD001; mTOR
MeSH Terms: conditions — Stomach Neoplasms | interventions — Everolimus

ARMS (1):
- RAD001 (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — 10 mg/day (2 tablets of 5 mg each)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of everolimus 10mg daily in patients with advanced gastric carcinoma (inoperable, recurrent or metastatic gastric cancer) whose cancer has progressed despite prior treatment.

ELIGIBILITY:
Inclusion criteria:

* Histological proven gastric adenocarcinoma
* Progressive disease during/ after prior treatment
* Treated with 1 or 2 chemotherapy regimen for advanced disease
* At least one measurable lesion by RECIST criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion criteria:

* History of another primary malignancy within 3 years
* Treated with 3 or more regimens for advanced gastric cancer
* Chronic treatment with steroids or another immunosuppressive agent
* A known history of HIV or hepatitis B seropositive, or active hepatitis C infection
* Patients with active, bleeding diathesis

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To Assess disease control rate (DCR) as defined CR + PR + SD assessed by RECIST criteria | 18 months

SECONDARY OUTCOMES:
Objective response rate (ORR) assessed by RECIST criteria | 18 months
To assess progression free survival (PFS) and overall survival (OS) | 18 months
To describe the safety profile (incidence and severity of adverse events, serious adverse events) assessed by NCI CTCAE version 3.0 | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Japan (8):
  - Novartis investigative Site, Aichi
  - Novartis investigative Site, Chiba
  - Novartis investigative Site, Ehime
  - Novartis Investigative Site, Hokkaido
  - Novartis investigative Site, Osaka
  - Novartis investigative Site, Shizuoka
  - Novartis Investigative Site, Tochigi
  - Novartis investigative Site, Tokyo

REFERENCES:
- [Result] Doi T, Muro K, Boku N, Yamada Y, Nishina T, Takiuchi H, Komatsu Y, Hamamoto Y, Ohno N, Fujita Y, Robson M, Ohtsu A. Multicenter phase II study of everolimus in patients with previously treated metastatic gastric cancer. J Clin Oncol. 2010 Apr 10;28(11):1904-10. doi: 10.1200/JCO.2009.26.2923. Epub 2010 Mar 15. PMID 20231677